CLINICAL TRIAL: NCT05164731
Title: Clinical Study of the Third Dose Immunization Schedule of COVID-19 Inactivated Vaccine, (Vero Cells) in Adults Aged 18 Years and Above After a Two-dose Schedule
Brief Title: Clinical Study of the Third Dose Immunization Schedule of COVID-19 Inactivated Vaccine, (Vero Cells) in Adults Aged 18 Years and Above
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Yunnan Center for Disease Control and Prevention (Other)
Responsible Party: Principal Investigator, Jingsi Yang, Senior Technologist, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20211102
Record Dates: First submitted 2021-12-14; First posted 2021-12-21 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: SARS-CoV2 Infection
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 3 months after two doses (Experimental): the third does was given 3 months after two doses
  Interventions: Biological: SARS-CoV-2 Vaccine, Inactivated (Vero Cell)
- 4 months after two doses (Experimental): the third does was given 4 months after two doses
  Interventions: Biological: SARS-CoV-2 Vaccine, Inactivated (Vero Cell)
- 5 months after two doses (Experimental): the third does was given 5 months after two doses
  Interventions: Biological: SARS-CoV-2 Vaccine, Inactivated (Vero Cell)
- 6 months after two doses (Experimental): the third does was given 6 months after two doses
  Interventions: Biological: SARS-CoV-2 Vaccine, Inactivated (Vero Cell)

INTERVENTIONS:
Biological: SARS-CoV-2 Vaccine, Inactivated (Vero Cell) — the third does was given 3, 4, 5 or 6 months after two doses

SUMMARY:
To evaluate the immunogenicity and safety of the third dose SARS-CoV-2 Vaccine, Inactivated (Vero Cell) in adults aged 18 years and above, who inoculated the third dose after 3, 4, 5, or 6 months since finished two doses schedule of Institute of Medical Biology Chinese Academy of Medical Sciences SARS-CoV-2 inactivated vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Axillary temperature ≤37.0 ℃.
2. aged 18 years and above, after 3, 4, 5, or 6 months since finished two doses schedule of Institute of Medical Biology Chinese Academy of Medical Sciences SARS-CoV-2 inactivated vaccine.
3. Proven legal identity, could come each visit.
4. Participants should understand the contents of the informed consent form, the vaccine in this trial, voluntarily sign the informed consent form.

Exclusion Criteria:

1. Persons with a clear history of SARS-CoV-2 infection.
2. Using blood products after basic immunization or receiving immunosuppressive therapy.
3. Participants who have a positive pregnancy test, or are breastfeeding, or plan to become pregnant, or plan to donate sperm or eggs from the screening to 6 months after vaccination.
4. Allergic to the active substance in the vaccine, any inactive substance or substance used in the preparation process (aluminum hydroxide, glycine);
5. History of abnormal clinical manifestations and serious diseases to be excluded, including but not limited to nervous system, cardiovascular system, blood and lymphatic system, immune system, kidney, liver, gastrointestinal tract, respiratory system, metabolism, bones and other system diseases, and a history of malignant tumors.
6. Diseases beyond drug control, such as high blood pressure, diabetes, asthma.
7. Those who developed acute disease within 2 weeks, or had symptoms of fever or upper respiratory tract infection within 7 days.
8. Immunization with any vaccine within 14 days.
9. Any other situations judged by investigators as not suitable for participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 880 (Estimated)
Dates: Start 2021-12-16 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Seroconversion rate of Neutralizing and IgG antibodies against SARS-CoV-2 | From 0 days to 6 month after the third dose
  Seroconversion rate of neutralizing antibodies and IgG against SARS-CoV-2 in serum for the third dose immunization schedule
SARS-CoV-2 specific memory B and T cell response | From 0 days to 6 month after the third dose
  SARS-CoV-2 specific memory B and T cell response for the third dose immunization schedule
Adverse reactions/events rate | 7 days after vaccination
  Occurence of adverse reactions/events after vaccination
Adverse reactions/events rate | 28 days after vaccination
  Occurence of adverse reactions/events after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zheng, Principal Investigator — Yunnan Center for Disease Control and Prevention
Locations (1):
- Mile City Centers for Disease Control and Prevention, Mile, Yunnan, China

IPD SHARING:
Plan to Share IPD: No